CLINICAL TRIAL: NCT00709150
Title: Multifaceted Depression Diabetes Program for Hispanics
Brief Title: Collaborative Depression Care Management in Treating Depressed Low-income Hispanics With Diabetes
Acronym: MDDP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH068468 (NIH); R01MH068468 (NIH); DSIR 82-SESQ
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2013-07

CONDITIONS: Depression
Keywords: Major Depression; Diabetes; Hispanics; Collaborative Depression Care Management
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients will receive collaborative depression care management.
  Interventions: Behavioral: Collaborative depression care management
- 2 (Active Comparator): Patients will receive enhanced usual care.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Collaborative depression care management — Collaborative depression care management will include acute depression treatment with antidepressant medication and/or counseling sessions based on structured problem solving therapy. Participants will also receive supportive patient navigation services and maintenance/relapse telephone monitoring. Counseling treatment will include 8 weekly 45-minute counseling sessions that are socio-culturally adaptated for the study population. The length of medication treatment will depend upon participants' severity of depression and may last up to 12 months.
  Arms: 1
Behavioral: Enhanced usual care — Participants will receive educational pamphlets on depression and a list of mental health resources in the community. Participants' primary care doctors will be free to prescribe antidepressant medication or provide other usual care.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of culturally adapted depression treatment for reducing depressive symptoms and improving adherence to diabetes self-care regimens in Hispanics with depression and diabetes.

DETAILED DESCRIPTION:
Diabetes, a disease in which the body does not properly produce or use insulin, is the fifth leading cause of death among Hispanics in the United States. The risk of comorbid depression among diabetics is twice as high as that of the general population, with depression rates among diabetic Hispanics as high as 33%. Symptoms of depression include feelings of sadness, anxiety, and guilt; lack of energy; changes in appetite; and lack of pleasure in previously enjoyed activities. These symptoms can make maintaining good diabetic management and self-care regimens difficult. Fortunately, depression is treatable with forms of psychotherapy and antidepressant medications. However, depression treatment adherence and response rates among the Hispanic population, especially among Hispanics of low socio-economic status, are lower than those of the general population. Depression treatment that is specifically adapted for the Hispanic culture may be best at helping diabetic Hispanics stick to their treatment and self-care plans. This study will evaluate the effectiveness of culturally adapted depression treatment for reducing depressive symptoms and improving adherence to diabetes self-care regimens in low-income Hispanics with depression and diabetes.

Participation in this study will last 18 months. All participants will first undergo baseline assessments that will include a 40-minute interview about personal health and feelings. Eligible participants will then be assigned randomly to receive either collaborative depression care management or enhanced usual care.

Participants assigned to receive collaborative depression care management will first be provided with information about depression treatment. Participants will then have the option of choosing between two depression treatments: counseling or antidepressant medications. Participants who choose to receive treatment with counseling will receive eight weekly 45-minute counseling sessions, conducted either on the phone or at the clinic. During these sessions, participants will undergo structured problem solving therapy (PST) and will learn strategies to manage their depressive symptoms. Participants who choose to receive treatment with antidepressant medication will be prescribed medication by a study doctor and will be monitored for any side effects throughout treatment. Medication treatment may last up to 12 months but will depend upon participants' severity of depression. After completing medication treatment, participants will be offered PST counseling. All participants receiving collaborative depression care management will also receive supportive patient navigation services and maintenance/relapse telephone monitoring.

Participants assigned to enhanced usual care will receive an educational pamphlet on depression and a list of mental health resources in the community. Participants' primary care doctors will be free to prescribe antidepressant medication or provide other usual care. All participants will undergo follow-up phone interviews about their status at Months 6, 12, and 18.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for major depression based on a score of greater than 2 for five or more symptoms, including one of the two cardinal depression symptoms and a nine-item depression scale of the Patient Health Questionnaire (PHQ-9) score of greater than 10
* Patient with diabetes
* Has attended two community safety net clinics

Exclusion Criteria:

* Current suicidal ideation
* Score of 8 or greater on the Alcohol Use Disorders Identification Test (AUDIT)
* Recent use of lithium or antipsychotic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2005-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Reduction in symptoms of major depression | Measured at Months 12, 18, and 24

SECONDARY OUTCOMES:
Quality of life | Measured at Months 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R. Ell, DSW, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California School of Social Work, Los Angeles, California, United States

REFERENCES:
- [Derived] Ell K, Katon W, Lee PJ, Kapetanovic S, Guterman J, Xie B, Chou CP. Depressive symptom deterioration among predominantly Hispanic diabetes patients in safety net care. Psychosomatics. 2012 Jul-Aug;53(4):347-55. doi: 10.1016/j.psym.2011.12.009. Epub 2012 Mar 27. PMID 22458987
- [Derived] Hay JW, Katon WJ, Ell K, Lee PJ, Guterman JJ. Cost-effectiveness analysis of collaborative care management of major depression among low-income, predominantly Hispanics with diabetes. Value Health. 2012 Mar-Apr;15(2):249-54. doi: 10.1016/j.jval.2011.09.008. Epub 2011 Dec 15. PMID 22433755
- [Derived] Ell K, Katon W, Xie B, Lee PJ, Kapetanovic S, Guterman J, Chou CP. One-year postcollaborative depression care trial outcomes among predominantly Hispanic diabetes safety net patients. Gen Hosp Psychiatry. 2011 Sep-Oct;33(5):436-42. doi: 10.1016/j.genhosppsych.2011.05.018. Epub 2011 Jul 19. PMID 21774987